CLINICAL TRIAL: NCT07380113
Title: An Exploratory Study Comparing Anrikefon With Nalfurafine in Improving Sleep Quality Among CKD-aP Patients Undergoing Hemodialysis: An Open-Label Randomized Controlled Clinical Trial
Brief Title: Anrikefon vs Nalfurafine for Sleep Quality in Hemodialysis Patients With CKD-aP
Acronym: Anrikefon
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Fengxian Li, Chief Physician, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-496-01
Record Dates: First submitted 2026-01-14; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pruritus Chronic; Kidney Diseases, Chronic; Renal Insufficiency, Chronic; Uremia; Chronic; Pruritus Due to Systemic Disorder (Disorder); Pruritus Due to Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Uremia; Bronchiolitis Obliterans Syndrome | interventions — TRK 820

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anrikefon (Experimental): Participants receive anrikefon injection at a dose of 0.3 μg/kg, administered three times per week after dialysis, for 4 consecutive weeks.
  Interventions: Drug: Anrikefon
- Nalfurafine (Active Comparator): Participants receive nalfurafine hydrochloride orally disintegrating tablets at a dose of 2.5 μg per day, administered orally after dinner, for 4 weeks.
  Interventions: Drug: Nalfurafine

INTERVENTIONS:
Drug: Anrikefon — intravenous administration
  Other Names: HSK21542
  Arms: Anrikefon
Drug: Nalfurafine — oral administration
  Other Names: TRK-820; Nalfurafine hydrochloride
  Arms: Nalfurafine

SUMMARY:
The goal of this clinical trial is to compare a new intravenous drug, Anruikefen, with a traditional oral medication, nalfurafine orally disintegrating tablets, in improving sleep quality in patients with chronic kidney disease-associated pruritus. Sleep quality will be primarily assessed using the Pittsburgh Sleep Quality Index (PSQI). The study will also evaluate the safety of Anruikefen.

The main questions it aims to answer are:

* Does Anruikefen injection improve sleep quality better than oral nalfurafine?
* Does Anruikefen injection improve patients' quality of life more than oral nalfurafine? Researchers will compare Anruikefen with nalfurafine (an active control drug) to evaluate differences in their effects on sleep quality in patients with chronic kidney disease-associated pruritus.

Participants will:

* Receive either Anruikefen injection (0.3 μg/kg, three times per week) or nalfurafine hydrochloride orally disintegrating tablets (2.5 μg once daily).
* Continue treatment for 4 weeks, followed by a 1-week safety follow-up.
* Complete the Pittsburgh Sleep Quality Index and other quality-of-life questionnaires after one month.

DETAILED DESCRIPTION:
This study adopts an open-label, randomized controlled design and enrolls patients with CKD-associated pruritus (CKD-aP) with a WI-NRS score ≥4. Participants are randomized to receive either anrikefon intravenous injection (0.3 μg/kg, three times per week) or nalfurafine orally disintegrating tablets administered orally (2.5 μg/day) for 4 weeks. The primary endpoint is the difference in sleep quality improvement assessed by the Pittsburgh Sleep Quality Index (PSQI). Secondary endpoints include Skindex-10, the 5-D Itch Scale, WI-NRS, KDQOL-36, Patient Global Impression of Change (PGIC), mechanical pain threshold, and serum proteomic analyses. Vital signs, laboratory parameters, and adverse events are monitored throughout the study to comprehensively evaluate the efficacy and safety of the two κ-opioid receptor agonist therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand the procedures and methods of this trial, be willing to strictly follow the clinical research protocol to complete this trial, and voluntarily sign the informed consent form.
2. Male or female individuals aged 18 or above and 75 or above.
3. Patients with end-stage renal disease received regular hemodialysis three times a week before the screening period (whether they met the requirements for regular dialysis was determined based on the opinions of the researchers).
4. Meet the diagnostic criteria for chronic kidney disease-associated pruritus (CKD-aP).

   1. Patients with chronic kidney disease (CKD) presenting with pruritus, with other identifiable causes of pruritus excluded.
   2. Pruritus occurring on at least 3 days within a 2-week period, with multiple episodes per day, each lasting for several minutes, and having an impact on the patient's daily life.
   3. Recurrent pruritus persisting for at least 6 weeks.A diagnosis requires that all three criteria above be met simultaneously.
5. The subjects were evaluated using the Worst Itch Numerical Rating Scale (WI-NRS) for the most severe pruritus intensity and met the baseline pruritus intensity of ≥ 4 points.

Exclusion Criteria:

1. Participants with other serious systemic diseases that may affect their ability to participate in the study, as assessed by the investigator, including but not limited to:

   1. Severe cardiovascular diseases, such as unstable angina, myocardial infarction, severe arrhythmias, World Health Organization (WHO) heart function classification III-IV during screening, poorly controlled hypertension or hypotension despite active treatment, and recurrent asthma.
   2. A history of cerebrovascular accident (CVA) within the last 6 months.
   3. Malignant tumors, excluding those that are curable, such as cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma of the skin, or any other cancer that has been cured (with no evidence of disease recurrence for 5 years).
2. It is expected to undergo kidney transplantation and/or parathyroidectomy during the study period.
3. The subjects are currently undergoing ultraviolet B treatment or are expected to receive such treatment during the study period.
4. Have participated in any clinical trials of other drugs or medical devices within one month prior to screening (treatment with drugs or medical devices that have received clinical trials).
5. Patients who have used the following drugs within 7 days before screening:

   1. those who have used opioids.
   2. those who must use opioids other than the investigational drug during the study period.
   3. those who has used gabapentin, pregabalin and calcineurin inhibitors;
   4. those who use drugs that can affect the efficacy judgment of anti-itching, including but not limited to antipsychotic drugs, sedative-hypnotic drugs, selective serotonin reuptake inhibitors (SSRIs), anti-anxiety drugs, or tricyclic antidepressants.
6. After screening and enrollment, new antihistamines (such as antihistamines and corticosteroids, etc. (oral, intravenous or topical)) were prescribed, or the types, dosages or frequencies of these drugs were changed.
7. There is a history of allergy to opioid drugs, or it is known that there is a history of allergy to investigatory drugs or components of remedial drugs or other drugs or excipients with similar chemical structures.
8. Severe hematological and liver function abnormalities during screening, meeting any one of the following clinical laboratory test results:

   1. Hematology: Hemoglobin < 80g/L.
   2. Liver function:

      * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5× upper limit of normal (ULN).
      * Total bilirubin (TBIL) > 2×ULN.
9. Subjects who had any active infections during screening and whom the researchers considered unsuitable for inclusion (including but not limited to acute hepatitis, skin infections, etc.).
10. As determined by the researchers, any other physical or mental illness or condition that may increase the risk of the trial, affect the subjects' compliance with the protocol, or affect the subjects' completion of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline, 4 weeks after medication
  Questionnaire survey

SECONDARY OUTCOMES:
5D-itching scale | Baseline，2/4 weeks after medication
  Questionnaire survey
Skindex-10 scale | Baseline，1 /2 /3/ 4 weeks after medication
  Questionnaire survey
WI-NRS score | Baseline, every dialysis day during the treatment period
  Questionnaire survey
Kidney Disease Quality of Life instrument™ - 36 items | Baseline, 4 weeks after medication
  Questionnaire survey
Patient Global Impression of Change | 4 weeks after medication
  Questionnaire survey
Mechanical pain threshold | Baseline, 4 weeks after medication
  The electronic pressure sensor pain measurement method involves connecting a probe with a relatively thin tip to a force sensor. Based on the principle of Newton's third law, it records in real time the magnitude of the force applied by the probe to the pain measurement site. The pressure number at which the subject first feels pain is the pain threshold.
Peripheral blood metabolomics analysis | Baseline, 4 weeks after medication
  Peripheral blood samples will be analyzed using liquid chromatography/mass spectrometry.
Peripheral blood proteomics analysis | Baseline, 4 weeks after medication
  The proteins in blood will be digested with trypsin to obtain peptides. The peptides will be analyzed by liquid nanochromatography coupled to mass spectrometry. The identification of the proteins will be carried out using the UniProt Homo Sapiens database using the Proteome Discoverer software (ThermoFisher Scientific).
  All proteomic markers in capillary blood will be reported in arbitrary units as a relative unit of measurement.